CLINICAL TRIAL: NCT06982079
Title: Effects of Sodium-Glucose Cotransporter 2 Inhibitors on Kidney Function in Advanced Chronic Kidney Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD102/2025
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease Stage 5; CKD Stage 4
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Eligible patients will receive dapagliflozin 10 mg in addition to standard of care
  Interventions: Drug: Dapagliflozin 10 mg
- Control arm (No Intervention): Eligible patients will receive standard of care only

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Dapagliflozin 10 mg will be added in addition to standard of care
  Arms: Dapagliflozin

SUMMARY:
The goal of this clinical trial is to evaluate whether dapagliflozin can reduce the risk of worsening kidney function or death from cardiovascular or renal causes in adults with advanced chronic kidney disease (CKD), with or without type 2 diabetes. The main questions it aims to answer are:

1. Does dapagliflozin reduce the rate of decline in kidney function or progression to end-stage kidney disease in adults with advanced CKD?
2. Does dapagliflozin reduce the risk of death from cardiovascular or renal causes in patients with advanced CKD?

Researchers will compare dapagliflozin to a placebo to see if dapagliflozin improves kidney and cardiovascular outcomes in this high-risk population.

DETAILED DESCRIPTION:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors, originally developed as oral antihyperglycemic agents for managing type 2 diabetes, have quickly gained recognition for their broad therapeutic benefits beyond glycemic control. Since their clinical introduction in 2012, SGLT2 inhibitors have demonstrated significant renoprotective and cardioprotective effects, reshaping treatment approaches in nephrology and cardiology.

Although these drugs have shown great promise, major clinical trials have typically excluded patients with advanced chronic kidney disease (CKD) (eGFR < 20 mL/min/1.73m²), those already on dialysis, and kidney transplant recipients-populations at the highest risk of kidney failure, cardiovascular complications, and mortality. This exclusion has left a critical gap in understanding the full potential of SGLT2 inhibitors in the most vulnerable patients. As such, current KDIGO guidelines have not recommended initiating SGLT2 inhibitors in patients with eGFR < 20 mL/min/1.73m².

CKD is a global health crisis, affecting approximately 10% of adults worldwide, with prevalence rising in Egypt, where 13% of adults are affected, especially in underserved rural areas. By 2040, CKD is projected to become the fifth leading cause of death worldwide.

For patients with kidney failure, the primary treatment options are renal replacement therapies like dialysis or transplantation. However, due to the scarcity of donor kidneys and the frequent presence of comorbidities in older populations, transplantation is often unfeasible. Consequently, most end-stage kidney disease (ESKD) patients rely on dialysis, a therapy that significantly lowers quality of life and increases mortality risk.

Preserving kidney function is a critical goal in CKD management, which is closely linked to better patient outcome. Incremental dialysis, a strategy aimed at preserving residual kidney function (RKF), shows promise but lacks robust clinical validation. Increasing evidence suggests that SGLT2 inhibitors, even in patients with advanced CKD, may offer significant reno- and cardioprotective benefits, reinforcing the need for further research into their efficacy in this population.

For instance, in the DAPA-CKD trial, which included patients with an eGFR as low as 25 mL/min/1.73m², dapagliflozin demonstrated a consistent reduction in cardiovascular and renal outcomes, even in those with severely impaired kidney function. A subgroup analysis of the DAPA-CKD trial comparing 624 patients with an eGFR <30 mL/min/1.73m2 to the remainder of the trial population with better kidney function, demonstrated that the efficacy of dapagliflozin in reducing cardiovascular and renal outcomes persisted in the population with impaired kidney function. Remarkably, patients who initiated dialysis during the trial continued to receive dapagliflozin or placebo, and those treated with dapagliflozin experienced a 21% reduction in relative risk for mortality. These findings challenge the traditional boundaries of SGLT2 inhibitor use, indicating potential benefits even in populations previously excluded from major trials.

Recent findings from the DAPA advKD trial (NCT05196347) further support this potential: in 180 patients with CKD stages 4-5 (eGFR 10-30 mL/min/1.73m²), dapagliflozin significantly slowed eGFR decline (-2.24 vs. -3.67 mL/min/1.73m²/yr in controls, p=0.019) and reduced composite renal outcomes (HR 0.50, p=0.019) over 1.6 years, despite a higher incidence of transient eGFR dips in the treatment group.

The 2023 UK Kidney Association Clinical Practice Guideline reinforces this paradigm shift, issuing a Grade 2B recommendation to consider SGLT2 inhibitor initiation in patients with eGFR <20 mL/min/1.73m² to slow disease progression. This guidance is supported by indirect evidence from trials continuing SGLT2 inhibition until kidney replacement therapy initiation, as well as EMPA-KIDNEY data showing unattenuated renal benefits down to eGFR 15 mL/min/1.73m².

Emerging clinical data further supports the efficacy of SGLT2 inhibitors in preserving RKF in patients undergoing dialysis. Recent case series have shown promising results, such as significant improvements in residual kidney urea clearance and reduced proteinuria among patients undergoing incremental hemodialysis while receiving SGLT2 inhibitors. Similarly, in patients on peritoneal dialysis, SGLT2 inhibitors have been effective in preserving RKF. Pharmacokinetic data also suggest that dapagliflozin is well tolerated, minimally dialyzable, and exhibits non-accumulating pharmacokinetic properties in patients on dialysis.

Given the substantial benefits of SGLT2 inhibitors in patients with less severe CKD, coupled with preliminary evidence suggesting their potential in advanced CKD and dialysis populations, there is a pressing need to explore their long-term efficacy and safety in these high-risk groups. This research aims to fill that gap, with the potential to redefine CKD management and offer new hope to patients facing the highest risks of poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged eighteen or older.
* Patients with advanced chronic kidney disease (i.e., eGFR < 20 mL/min/1.73m2)not on dialysis

Exclusion Criteria:

* Autosomal dominant polycystic kidney disease (ADPKD).
* Type 1 diabetes mellitus
* Patients on SGLT2 inhibitors.
* History of ketoacidosis in the last 3 months.
* Known hypersensitivity to SGLT2 inhibitors.
* Known hepatic impairment.
* Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in the eGFR slope | 1 year
  To determine whether dapagliflozin is superior to standard of care only in reducing the eGFR slope.
Time to start of renal replacement therapy | 1 year
  Kidney failure is defined as need for renal replacement therapy either by hemodialysis or kidney transplant

SECONDARY OUTCOMES:
Incidence of hospitalization for heart failure | 1 year
  To determine if dapagliflozin is superior to standard of care only in reducing the incidence of heart failure
Number of participants with all-cause mortality | 1 year
  To determine whether dapagliflozin is superior to standard of care only in reducing all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD Work Group. KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney Int. 2024 Apr;105(4S):S117-S314. doi: 10.1016/j.kint.2023.10.018. No abstract available. PMID 38490803
- [Background] Roddick AJ, Wonnacott A, Webb D, Watt A, Watson MA, Staplin N, Riding A, Lioudaki E, Kuverji A, Kossi ME, Holmes P, Holloway M, Fraser D, Carvalho C, Burton JO, Bhandari S, Herrington WG, Frankel AH. UK Kidney Association Clinical Practice Guideline: Sodium-Glucose Co-transporter-2 (SGLT-2) Inhibition in Adults with Kidney Disease 2023 UPDATE. BMC Nephrol. 2023 Oct 25;24(1):310. doi: 10.1186/s12882-023-03339-3. PMID 37880609
- [Background] Moral Berrio E, De La Flor JC, Arambarri Segura M, Rodriguez-Doyaguez P, Martinez Calero A, Zamora R, Cieza-Terrones M, Yuste-Lozano C, Sanchez de la Nieta Garcia MD, Nieto Iglesias J, Vozmediano Poyatos C. Effects of Sodium-Glucose Cotransporter 2 Inhibitors in Diabetic and Non-Diabetic Patients with Advanced Chronic Kidney Disease in Peritoneal Dialysis on Residual Kidney Function: In Real-World Data. Medicina (Kaunas). 2024 Jul 24;60(8):1198. doi: 10.3390/medicina60081198. PMID 39202480
- [Background] Levey AS, Gansevoort RT, Coresh J, Inker LA, Heerspink HL, Grams ME, Greene T, Tighiouart H, Matsushita K, Ballew SH, Sang Y, Vonesh E, Ying J, Manley T, de Zeeuw D, Eckardt KU, Levin A, Perkovic V, Zhang L, Willis K. Change in Albuminuria and GFR as End Points for Clinical Trials in Early Stages of CKD: A Scientific Workshop Sponsored by the National Kidney Foundation in Collaboration With the US Food and Drug Administration and European Medicines Agency. Am J Kidney Dis. 2020 Jan;75(1):84-104. doi: 10.1053/j.ajkd.2019.06.009. Epub 2019 Aug 28. PMID 31473020
- [Background] Kalantar-Zadeh K, Jafar TH, Nitsch D, Neuen BL, Perkovic V. Chronic kidney disease. Lancet. 2021 Aug 28;398(10302):786-802. doi: 10.1016/S0140-6736(21)00519-5. Epub 2021 Jun 24. PMID 34175022
- [Background] Inker LA, Eneanya ND, Coresh J, Tighiouart H, Wang D, Sang Y, Crews DC, Doria A, Estrella MM, Froissart M, Grams ME, Greene T, Grubb A, Gudnason V, Gutierrez OM, Kalil R, Karger AB, Mauer M, Navis G, Nelson RG, Poggio ED, Rodby R, Rossing P, Rule AD, Selvin E, Seegmiller JC, Shlipak MG, Torres VE, Yang W, Ballew SH, Couture SJ, Powe NR, Levey AS; Chronic Kidney Disease Epidemiology Collaboration. New Creatinine- and Cystatin C-Based Equations to Estimate GFR without Race. N Engl J Med. 2021 Nov 4;385(19):1737-1749. doi: 10.1056/NEJMoa2102953. Epub 2021 Sep 23. PMID 34554658
- [Background] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Background] Heerspink HJL, Sjostrom CD, Jongs N, Chertow GM, Kosiborod M, Hou FF, McMurray JJV, Rossing P, Correa-Rotter R, Kurlyandskaya R, Stefansson BV, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Effects of dapagliflozin on mortality in patients with chronic kidney disease: a pre-specified analysis from the DAPA-CKD randomized controlled trial. Eur Heart J. 2021 Mar 31;42(13):1216-1227. doi: 10.1093/eurheartj/ehab094. PMID 33792669
- [Background] Foreman KJ, Marquez N, Dolgert A, Fukutaki K, Fullman N, McGaughey M, Pletcher MA, Smith AE, Tang K, Yuan CW, Brown JC, Friedman J, He J, Heuton KR, Holmberg M, Patel DJ, Reidy P, Carter A, Cercy K, Chapin A, Douwes-Schultz D, Frank T, Goettsch F, Liu PY, Nandakumar V, Reitsma MB, Reuter V, Sadat N, Sorensen RJD, Srinivasan V, Updike RL, York H, Lopez AD, Lozano R, Lim SS, Mokdad AH, Vollset SE, Murray CJL. Forecasting life expectancy, years of life lost, and all-cause and cause-specific mortality for 250 causes of death: reference and alternative scenarios for 2016-40 for 195 countries and territories. Lancet. 2018 Nov 10;392(10159):2052-2090. doi: 10.1016/S0140-6736(18)31694-5. Epub 2018 Oct 16. PMID 30340847
- [Background] Dobre M. Safety of SGLT2 Inhibitors in CKD: Walking the Fine Line. Clin J Am Soc Nephrol. 2022 Jun;17(6):774-776. doi: 10.2215/CJN.04900422. Epub 2022 May 26. No abstract available. PMID 35618341
- [Background] De La Flor JC, Villa D, Cruzado L, Apaza J, Valga F, Zamora R, Marschall A, Cieza M, Deira J, Rodeles M. Efficacy and Safety of the Use of SGLT2 Inhibitors in Patients on Incremental Hemodialysis: Maximizing Residual Renal Function, Is There a Role for SGLT2 Inhibitors? Biomedicines. 2023 Jul 6;11(7):1908. doi: 10.3390/biomedicines11071908. PMID 37509547
- [Background] Chertow GM, Vart P, Jongs N, Toto RD, Gorriz JL, Hou FF, McMurray JJV, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Langkilde AM, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effects of Dapagliflozin in Stage 4 Chronic Kidney Disease. J Am Soc Nephrol. 2021 Sep;32(9):2352-2361. doi: 10.1681/ASN.2021020167. Epub 2021 Jul 16. PMID 34272327
- [Background] Barreto J, Borges C, Rodrigues TB, Jesus DC, Campos-Staffico AM, Nadruz W, Luiz da Costa J, Bueno de Oliveira R, Sposito AC. Pharmacokinetic Properties of Dapagliflozin in Hemodialysis and Peritoneal Dialysis Patients. Clin J Am Soc Nephrol. 2023 Aug 1;18(8):1051-1058. doi: 10.2215/CJN.0000000000000196. Epub 2023 May 25. PMID 37227937